CLINICAL TRIAL: NCT00209456
Title: GEHC Has Decided Not to Provide This Detail But Will Rely on the Brief Title
Brief Title: Dopamine Transporter Scintigraphy Imaging (DAT-Imaging) in Patients With Lewy Body Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PDT301
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Lewy Body Dementia; Non-DLB Dementia; Alzheimer's; Vascular Dementia
Keywords: Lewy Body Dementia; non-DLB dementia; Dopamine Transporter; Striatal Uptake
MeSH Terms: conditions — Lewy Body Disease; Dementia, Vascular | interventions — ioflupane

INTERVENTIONS:
Drug: DatSCAN

SUMMARY:
The study is designed to determine the diagnostic efficacy of the visual assessment of SPECT scans in differentiating between probable dementia with Lewy Bodies (DLB) and non-DLB dementia subjects determined by the clinical diagnosis of an independent expert consensus panel used as the standard of truth.

DETAILED DESCRIPTION:
GEHC had decided notto provide this detail

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adults between 55 to 90 years of age with an established diagnosis for dementia in accordance with DSM-IV criteria and have to fulfil at least one of the following: The ICC criteria for probable and possible DLB, the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer Disease and Related Disorders Association (NINCDS-ADRDA) for Alzheimer's Disease (AD), or the National Institute of Neurological and Communicative Disorders and Association Internationale Pour la Recherche et l'Enseignement en Neurosciences (NINCS-AIREN) for Vascular Dementia (VaD).

Exclusion Criteria:

* Subjects are not eligible if they have a Mini Mental State Examination (MMSE) score of <10 and use medication known or suspected to interact with the striatal uptake DaTSCAN to the dopamine transporter.
* Furthermore subjects are not eligible if they were diagnosed with idiopathic Parkinson's Disease (PD), with persistent severe depression, normal pressure hydrocephalus, multiple system atrophy, cortico-basal degeneration or Huntington's Chorea Disease.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326
Dates: Start 2003-11

PRIMARY OUTCOMES:
Sensitivity and specificity of DaTSCAN SPECT scans in differentiating between probable dementia with Lewy Bodies (DLB) and non-DLB dementia subjects.

SECONDARY OUTCOMES:
Accuracy, positive predictive value and negative predictive value of DaTSCAN SPECT
Semi-quantitative analysis of the striatal uptake ratios of DaTSCAN SPECT images.
Impact of DaTSCAN SPECT analysis on the confidence of diagnosis.
Findings in relation to probable, possible and no-DLB.
Efficacy analysis at 12-month follow-up period.
Safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pignot, PhD, Study Director — GE Healthcare
Locations (1):
- Amersham Buchler GmbH Co. KG, Ismaning, Germany

REFERENCES:
- [Derived] O'Brien JT, Oertel WH, McKeith IG, Grosset DG, Walker Z, Tatsch K, Tolosa E, Sherwin PF, Grachev ID. Is ioflupane I123 injection diagnostically effective in patients with movement disorders and dementia? Pooled analysis of four clinical trials. BMJ Open. 2014 Jul 3;4(7):e005122. doi: 10.1136/bmjopen-2014-005122. PMID 24993764